CLINICAL TRIAL: NCT00619164
Title: A Double-Blind Study of E5555 in Japanese Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E5555-J081-207
Record Dates: First submitted 2007-12-05; First posted 2008-02-20 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2010-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Platelet Aggregation Inhibitors; Coronary Stenosis; Coronary Thrombosis
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Stenosis; Coronary Thrombosis | interventions — E 5555

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: E5555
- 2 (Experimental)
  Interventions: Drug: E5555
- 3 (Experimental)
  Interventions: Drug: E5555
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E5555 — E5555, 50 mg (tablet), taken orally, once a day.
  Arms: 1
Drug: E5555 — E5555, 100 mg (tablet), taken orally, once a day.
  Arms: 2
Drug: E5555 — E5555, 200 mg (tablet), taken orally, once a day.
  Arms: 3
Drug: Placebo — Placebo tablet taken orally, once a day.
  Arms: 4

SUMMARY:
The purpose of this study is to assess the safety and tolerability of E5555 in Japanese patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. 45 - 80 years old (at time of informed consent)
2. Male or female (females of childbearing potential must be contracepted)
3. Confirmed acute coronary syndrome

Exclusion Criteria:

1. Unwilling or unable to provide informed consent
2. History of acquired or congenital bleeding disorder, coagulopathy, or platelet disorder
3. Recent trauma or major surgery
4. Evidence of active pathological bleeding at screening or history of gastrointestinal or genitourinary bleeding with unknown cause within 24 weeks prior to screening
5. History of intracranial bleeding or history of hemorrhagic retinopathy
6. History of New York Heart Association (NYHA) class III or IV congestive heart failure
7. Pregnant or lactating women

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events, bleeding events, clinical laboratory tests, Coagulation tests, vital signs and 12-lead ECG. | 3 months

SECONDARY OUTCOMES:
Major cardiac adverse events, biomarkers, platelet aggregation inhibition, plasma concentration. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Masaru Takeuchi, Study Director — New Product Development, Clinical Research Center, Eisai Co., Ltd.
Locations (33):
- Japan (33):
  - Toyoake, Aichi-ken
  - Fukuoka, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Gifu, Gifu
  - Ōgaki, Gifu
  - Fukuyama, Hiroshima
  - Higashi-Hiroshima, Hiroshima
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Amagasaki, Hyōgo
  - Himaji, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Kagoshima, Kagoshima-ken
  - Yokohama, Kanagawa
  - Ōmura, Nakasaki
  - Beppu, Oita Prefecture
  - Urazoe, Okinawa
  - Osaka, Osaka
  - Wako, Saitama
  - Komatsushimachō, Tokushima
  - Bunkyo, Tokyo
  - Fuchū, Tokyo
  - Hachiōji, Tokyo
  - Kodaira, Tokyo
  - Nerima City, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku, Tokyo
  - tabashi City, Tokyo
  - Tanabe, Wakayama